CLINICAL TRIAL: NCT06587776
Title: Investigation of the Regulation of Retinal and Choroidal Blood Vessels in Various Ocular Axes Lengths Based on Ultra-widefield Swept-source Optical Coherence Tomography Angiography Detection With Changes in Body Position
Brief Title: Investigation of the Regulation of Retinal and Choroidal Blood Vessels in Various AL Based on WF SS-OCTA Detection With Changes in Body Position
Status: Not yet recruiting | Type: Observational
Sponsor: Science and Technology Department of Sichuan Province (Other)
Responsible Party: Sponsor
Other Study IDs: YH-EC-SOP-019(F)-001
Record Dates: First submitted 2024-09-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal axial length grooup: At the screening stage, the axial length of the subjects was measured by IOL master 700. If the other conditions were met, the subjects would be included in this group If the axial length is between 23mm and 24mm.
- Long axial group: At the screening stage, the axial length of the subjects was measured by IOL master 700. If the other conditions were met, the subjects would be included in this group if the axial length is greater than 24mm.

SUMMARY:
This prospective observational study aims to understand the effects of different subaxial body positions on choroidal and retinal blood vessel density. The main questions it aims to answer are as follows:1) How do retinal and choroidal blood vessels adjust and repair after changes in body position?2) Is the change of body position related to the factors that cause myopia？ 3) Are there any differences in the regulation ability of fundus blood vessels in people with different ocular axes under the condition of changes in body position?

DETAILED DESCRIPTION:
This project will use the wide field swept-source optical coherence tomography angiography, combined with data analysis and mining methods, to explore the self-adjustment and change mode and mechanism of retinal and choroidal blood vessels in the case of posture changes in an all-round and multi-angle way. There would be three kinds of postural changes, one is 15° head-up position, one is supine position, and the other is 15° head-down position. Relevant ophthalmological measurements would be performed before and after the postural changes. The objective is to discover the three-dimensional change mode of retinal and choroid blood vessels in different postures and compare the differences among people with different lengths of ocular axes, and to elucidate the relationship between the mode and ability of retinal and choroidal blood vessels to adjust and repair changes after changes in body position and myopia, to provide more ideas and objective basis for the occurrence and development of myopia, and lay a foundation for further research. It is of great significance to innovate the pathogenesis of myopia, deepen the theoretical understanding, and guide the prevention and control of myopia.

ELIGIBILITY:
Inclusion Criteria:

1. Corrected visual acuity ≥1.0 (international standard visual acuity chart);
2. Age 10-40 years old;
3. In good health;
4. Give informed consent and volunteer for the study. The process of obtaining informed consent complies with GCP regulations.

Exclusion Criteria:

1. Can not cooperate with the completion of relevant inspection and data collection;
2. Pregnant and lactating women;
3. Patients with amblyopia, glaucoma, retinitis pigmentosa, senile macular degeneration, retinal artery obstruction, retinal vein obstruction, diabetic retinopathy and other eye diseases that may affect the blood circulation and vascular diameter of the retina and vein, or those who have undergone intraocular surgery;
4. Patients with cardiovascular and cerebrovascular diseases, endocrine diseases, autoimmune diseases;
5. Long history of smoking and drinking;
6. History of ocular trauma;
7. The mentally ill;
8. Those who have taken drugs that affect blood circulation in the past 3 months;

Ages: 10 Years to 40 Years | Sex: All
Age Groups: Child, Adult
Study Population: Healthy people in Chengdu City will be recruited through advertisement, and those who meet the inclusion and exclusion criteria will enter the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Retinal blood flow density | During the procedure
  Two modes of SS-OCTA will be used for scanning, one is the wide-angle range of 24mm*20mm grid for quantitative analysis of choroidal and retinal vascular density. The other is a scanning range of 12mm*12mm mode, and the choroidal thickness, choroidal vascular volume ratio, and the area and perimeter of the macular avascular zone will be analysed.
Intraocular pressure | During the procedure
  iCare handheld contact tonometer wIll be used to measure the intraocular pressure of the subjects
Choroidal blood flow density | During the procedure
  Two modes of SS-OCTA will be used for scanning, one is the wide-angle range of 24mm*20mm grid for quantitative analysis of choroidal and retinal vascular density. The other is a scanning range of 12mm*12mm mode, and the choroidal thickness, choroidal vascular volume ratio, and the area and perimeter of the macular avascular zone will be analysed.
Choroidal thickness | During the procedure
  Two modes of SS-OCTA will be used for scanning, one is the wide-angle range of 24mm*20mm grid for quantitative analysis of choroidal and retinal vascular density. The other is a scanning range of 12mm*12mm mode, and the choroidal thickness, choroidal vascular volume ratio, and the area and perimeter of the macular avascular zone will be analysed.
Foveal avascular zone area | During the procedure
  Two modes of SS-OCTA will be used for scanning, one is the wide-angle range of 24mm*20mm grid for quantitative analysis of choroidal and retinal vascular density. The other is a scanning range of 12mm*12mm mode, and the choroidal thickness, choroidal vascular volume ratio, and the area and perimeter of the macular avascular zone will be analysed.

SECONDARY OUTCOMES:
Axial length | Baseline, pre-procedure
  IOL Master700 will be used for the acquisition of axial length data.

IPD SHARING:
Plan to Share IPD: No